CLINICAL TRIAL: NCT01234077
Title: A Single Blind Randomized Study Comparing In-laboratory Polysomnography Electrocardiogram to Simultaneously Recorded In-laboratory Electrocardiogram on the CPC M1 Device and Compared to Home Recorded Electrocardiogram With the CPC M1 Device.
Brief Title: Study Comparing In-laboratory Polysomnography Electrocardiogram (PSG ECG) to Simultaneously Recorded In-laboratory ECG on the CPC M1 Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: MyCardio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPC M1
Record Dates: First submitted 2010-10-29; First posted 2010-11-04 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Sleep Disorder
Keywords: scheduled for a polysomnogram (overnight sleep study)
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ECG recording (No Intervention): In-laboratory vs. in-home recordings
  Interventions: Device: CPC M1

INTERVENTIONS:
Device: CPC M1 — CPC M1
  Other Names: in-laboratory vs. in-home recordings

SUMMARY:
Research study that will test a portable device (CPC M1) that records: body movement; heart activity (ECG; snoring; and body position during sleep. The Food and Drug Administration (FDA) has not approved this device for use except in a research setting.

The purposes of this study are to: a) determine if the ECG data collected using the CPC M1 device is at least as good as the ECG data collected during a diagnostic, in-lab polysomnogram (PSG) (or sleep study) and b) determine if in-home monitoring with the device will provide similar results compared to an in-lab PSG.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (males and females) 18 to 70 years of age with a suspected sleep disorder.
2. Subjects or legal guardians are able to verbalize an understanding of the consent form, provide written informed consent, and verbalize willingness to complete study procedures.
3. Adequate dexterity to apply and remove the CPC M1 device.

Exclusion Criteria:

1. Patients with atrial fibrillation and ventricular tachycardia.
2. Patients with an inability to apply the CPC M1 device.
3. Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of an electrocardiogram-based method to predict the presence of a sleep disorder. | 6 months
  Does the ECG-based data obtained from a portable device correlate to a similar analysis of simultaneously recorded ECG data obtained from standard polysomnography?
Sensitivity and specificity of an electrocardiogram-based method to predict the presence of a sleep disorder. | 6 months
  What is the sensitivity/specificity of the ECG-based method recorded in-lab vs. in the home.

CONTACTS AND LOCATIONS:
Overall Officials: John Harrington, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Magnusdottir S, Hilmisson H. Ambulatory screening tool for sleep apnea: analyzing a single-lead electrocardiogram signal (ECG). Sleep Breath. 2018 May;22(2):421-429. doi: 10.1007/s11325-017-1566-6. Epub 2017 Sep 7. PMID 28884264
- [Derived] Harrington J, Schramm PJ, Davies CR, Lee-Chiong TL Jr. An electrocardiogram-based analysis evaluating sleep quality in patients with obstructive sleep apnea. Sleep Breath. 2013 Sep;17(3):1071-8. doi: 10.1007/s11325-013-0804-9. Epub 2013 Jan 25. PMID 23354509